CLINICAL TRIAL: NCT05951062
Title: Benefits of Patient-centered Medication Management Education on Blood Pressure and Health Outcomes for Hypertensive Elderly Patients in Residential Care Facility
Brief Title: Trans-theoretical Model Based Home Visiting on Medication Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Chang (Other)
Responsible Party: Sponsor-Investigator, Jing Chang, Director of Cadre Health Office, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-KY-143
Record Dates: First submitted 2023-06-20; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Medication Adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- five sessions of educational interview (Experimental): The intervention included five educational sessions focused on anti-hypertensive medication-related information, the importance of medication refills, motivation, self-management and self-check skills.
  Interventions: Behavioral: behavior management for anti-hypertensive medication
- treatment as usual (Other): usual care provided by facility,such as regular blood pressure checking and meals
  Interventions: Other: placebo group

INTERVENTIONS:
Behavioral: behavior management for anti-hypertensive medication — five sessions of educational interview and home visiting to improve medication-related self-management skills
  Arms: five sessions of educational interview
Other: placebo group — treatment as usual
  Arms: treatment as usual

SUMMARY:
This study was a single-blinded, two-armed, randomized controlled trial comparing a medication self-management intervention to usual care for hypertensive elderly in the residential care facility.

To explore the effect of stage-matched tailored education on disease management for hypertensive elderly. Patient were randomly assigned to either a 6-month trans-theoretical model-based medication management intervention group or a treatment-as-usual group. we would like to improve its adherence to the medicine prescribed by their own physician through five sessions of face-to-face interview which focused on anti-hypertensive medication-related information, the importance of medication refills, motivation, self-management and self-check skills.

DETAILED DESCRIPTION:
This study was a single-blinded, two-armed, randomized controlled trial comparing a medication self-management intervention to usual care for hypertensive elderly in the residential care facility. From October 2018 to November 2018, convenience sampling was used to recruit 120 participants from one of the most extensive facilities in Zhengzhou, China. Individuals aged 65 years of age or older diagnosed had stage I or stage II hypertension (140-159/90-99 mm Hg or 160-180/100-110 mm Hg, respectively), as confirmed by the professional physician and prescribed anti-hypertensive medication by the physician for at least six months and with an estimated life expectancy of no less than six months were included.The intervention included five educational sessions focused on anti-hypertensive medication-related information, the importance of medication refills, motivation, self-management and self-check skills.

ELIGIBILITY:
Inclusion Criteria:

1. aged 65 years of age or older
2. diagnosed with a stage I or stage II hypertension (140-159/90-99 mm Hg or 160-180/100-110 mm Hg, respectively), as confirmed by the professional physician
3. prescribed anti-hypertensive medication by the physician for at least six months

Exclusion Criteria

1. unable to communicate and take medications by themselves.
2. with an estimated life expectancy of no more than six months. -

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — >=65y
Enrollment: 120 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 0.3month.6month.3years
  Sphygmomanometers，assessing Change from Baseline Blood Pressure at 3 years

SECONDARY OUTCOMES:
medication adherence | 0.3month.6month.3years
  Adherence to Refills and Medications Scale，The raw scores are changed from original metric to a 10-40 metric, in which lower scores means higher level of adherence
medication self-efficiency | 0.3month.6month.3years
  Self-efficiency for appropriate medication use scale (SEAMS),It has 13 items and patients are asked about their level of confidence about taking medication correctly under a varied circumstance. Each item is evaluated by three-point Likert respond scale (1=not confident, 2=somewhat confident, 3=very confident), higher score means higher confidence
patient activation | 0.3month.6month.3years
  patient activation measure-10 (PAM-10) scale.The raw scores are changed from original metric to a 0-100 metric, in which higher scores means higher level of activation

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chang, Master, Study Director — The First Affiliated Hospital of Zhengzhou University，Zhengzhou,China. ZIP：450000; YiJing Chen, Master, Principal Investigator — Wuhan mental health center,Wuhan,China. ZIP：430000
Locations (1):
- Senior Residences of Henan Province, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make data available.